CLINICAL TRIAL: NCT06989359
Title: A Phase 2 Study to Assess ADX-038 in Participants With Complement-Mediated Kidney Disease
Brief Title: Phase 2 Study of ADX-038 in Complement-Mediated Kidney Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ADARx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADX-038-201
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: IgAN; C3G; Complement-mediated Kidney Disease; IgA Nephropathy (IgAN); IC-MPGN
Keywords: IgA Nephropathy; IgAN; C3G; IC-MPGN; complement-mediated kidney disease
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ADX-038 Dose Level 1 - IgAN (Experimental)
  Interventions: Drug: ADX-038 Dose Level 1
- ADX-038 Dose Level 1 - C3G (Experimental)
  Interventions: Drug: ADX-038 Dose Level 1
- ADX-038 Dose Level 2 - IgAN (Experimental)
  Interventions: Drug: ADX-038 Dose Level 2

INTERVENTIONS:
Drug: ADX-038 Dose Level 2 — siRNA duplex oligonucleotide
  Arms: ADX-038 Dose Level 2 - IgAN
Drug: ADX-038 Dose Level 1 — siRNA duplex oligonucleotide
  Arms: ADX-038 Dose Level 1 - C3G; ADX-038 Dose Level 1 - IgAN

SUMMARY:
This Phase 2 study is designed to assess the safety, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of ADX-038 in adults with complement-mediated kidney diseases.

ELIGIBILITY:
Inclusion Criteria:

* Mean eGFR
* Clinical evidence of active kidney disease
* Been on supportive care
* vaccine requirements
* Females must not be pregnant or breastfeeding
* Men must agree to use acceptable contraception and not donate sperm
* IgAN: confirmed disease by kidney biopsy performed within 60 months prior to screening
* C3G/IC-MPGN: confirmed disease by kidney biopsy performed within 18 months prior to screening

Exclusion Criteria:

* Hereditary or acquired complement deficiency
* Kidney transplant or renal replacement therapy
* History of solid organ transplant
* Other kidney disease
* History of recurrent invasive infections
* Received complement inhibitor treatments
* Active systemic viral, bacterial, or fungal infection
* Liver dysfunction
* No donating blood

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of ADX-038 | Length of study - 36 months
  Incidence and severity of TEAEs

CONTACTS AND LOCATIONS:
Overall Officials: Aditya Patel, MD, Study Director — ADARx Pharmaceuticals, Inc.
Locations (12):
- United States (5):
  - ADARx Clinical Site, Shreveport, Louisiana
  - ADARx Clinical Site, Shelby, Michigan
  - ADARx Clinical Site, Dakota Dunes, South Dakota
  - ADARx Clinical Site, Dallas, Texas
  - ADARx Clinical Site, Houston, Texas
- ADARx Clinical Site, Wollongong, New South Wales, Australia
- Hong Kong (2):
  - ADARx Clinical Site, Pok Fu Lam
  - ADARx Clinical Site, Shatin
- South Korea (4):
  - ADARx Clinical Site, Gyeonggi-do, New South Wales
  - ADARx Clinical Site, Seoul, New South Wales
  - ADARx Clinical Site, Cheonan
  - ADARx Clinical Site, Seoul

IPD SHARING:
Plan to Share IPD: Undecided